CLINICAL TRIAL: NCT00675675
Title: TRECC: Neurocognitive Correlates of Behavioral Treatment for Childhood Tic Disorders
Brief Title: Neurocognitive Correlates of Behavioral Treatment for Childhood Tic Disorders
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: John Piacentini (Other)
Responsible Party: Sponsor-Investigator, John Piacentini, Professor in Residence, University of California, Los Angeles
Organization: University of California, Los Angeles (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: UCLAP500772484; P50MH077248 (NIH)
Record Dates: First submitted 2008-05-07; First posted 2008-05-12 (Estimated); Last update posted 2015-08-21 (Estimated); Status verified 2015-08

CONDITIONS: Tic Disorder
Keywords: Tourette Syndrome; Chronic Tic Disorder; Tics; Behavior Therapy; Habit Reversal Training; Child; Adolescent; Neuroimaging
MeSH Terms: conditions — Tic Disorders; Tourette Syndrome; Tics

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Comprehensive Behavioral Intervention for Tics (CBIT) (Active Comparator): Habit Reversal Training (HRT) plus functional assessment/intervention designed to identify and ameliorate environmental triggers for and consequences to tics that might serve to maintain and/or generalize these symptoms
  Interventions: Behavioral: Comprehensive Behavioral Intervention for Tics (CBIT)
- Minimal Contact Waitlist (Other): Bimonthly phone check-in to assess illness severity and maximize subject retention
  Interventions: Behavioral: Minimal Contact Waitlist

INTERVENTIONS:
Behavioral: Comprehensive Behavioral Intervention for Tics (CBIT) — Habit Reversal Training plus functional assessment/intervention designed to identify and ameliorate tic triggers (antecedents) and maintaining consequences.
  Arms: Comprehensive Behavioral Intervention for Tics (CBIT)
Behavioral: Minimal Contact Waitlist — Bimonthly phone check-in to assess clinical status and enhance subject retention
  Arms: Minimal Contact Waitlist

SUMMARY:
The study aims to clarify the functional anatomy of key brain circuits associated with cognitive control in children and adolescents with chronic tic disorders (CTD) and to compare and contrast hypothesized mechanisms related to increased tic control associated with Habit Reversal Training, a behavioral treatment that been previously shown to be effective in treating CTD. We also seek to better understand the relationship between fMRI and quantitative EEG in relevant brain circuits with the hope of establishing EEG as a valid and cost-effective marker of treatment responsiveness. A total of 25 subjects will be randomized to 10 weeks of Habit Reversal Training (HRT), a behavioral treatment, and 25 to 10 weeks of minimal-contact waitlist. Treatment responders will be re-assessed at three months. Waitlist nonresponders will be provided with 10 weeks of HRT. Study assessments, including a neurocognitive battery and quantitative EEG will be administered at baseline, Wk 5, Wk 10, and 3-month follow-up. Neuroimaging (fMRI) will be conducted at baseline and Wk 10.

ELIGIBILITY:
Inclusion Criteria:

* DSM-IV diagnostic criteria for CTD (CMVT or TS)
* Clinical Global Impressions - Severity Score > 3 (moderately ill or worse)
* YGTSS Total Score > 14 (or Total Score > 10 if CTD with motor tics only)
* Unmedicated or on stable psychotropic medication for at least 6 weeks prior to study entry, with no planned changes for duration of study participation
* Child is fluent English speaker
* Parental Informed Consent and Child Informed Assent.

Exclusion Criteria:

* Total YGTSS Score>35 (Cases above this threshold otherwise eligible will be reviewed by Clinical Caseness Panel for potential study participation)
* IQ < 80 on the Wechsler Abbreviated Scale of Intelligence (WASI)
* Problematic Substance Use or DSM-IV Conduct Disorder in past 3 months
* Lifetime DSM-IV diagnosis of PDD, Mania, or Psychotic Disorder
* Any serious psychiatric, psychosocial, or neurological condition requiring immediate treatment other than that provided in the current study
* Previous treatment with four or more sessions of HRT for tics
* Contraindication to fMRI scan

Ages: 9 Years to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 53 (Actual)
Dates: Start 2007-07; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Clinical Global Impressions - Improvement | Wks 0, 5, 10

SECONDARY OUTCOMES:
Yale Global Tic Severity Scale | Wks 0, 5, 10

CONTACTS AND LOCATIONS:
Overall Officials: John Piacentini, Ph.D., Study Director — University of California, Los Angeles; James McCracken, M.D., Principal Investigator — University of California, Los Angeles
Locations (1):
- University of California, Los Angeles, Los Angeles, California, United States